CLINICAL TRIAL: NCT00089973
Title: Phase II, Open Label Study of Ispinesib in Subjects With Advanced or Metastatic Breast Cancer
Brief Title: Study Of Ispinesib In Subjects With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSP20001
Record Dates: First submitted 2004-08-18; First posted 2004-08-20 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2017-08

CONDITIONS: Neoplasms, Breast
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ispinesib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB-715992 (Experimental): Females with advanced or metastatic breast cancer were administered Ispinesib
  Interventions: Drug: Ispinesib

INTERVENTIONS:
Drug: Ispinesib — Given intravenously at a dose of 18 milligram (mg)/ meter square (m^2).

SUMMARY:
The purpose of this research study is to find how breast cancer responds to the investigational drug, Ispinesib. An investigational drug is a drug that has not been approved by the Food and Drug Administration (FDA) and is available for research use only. In particular, this study will try is to find the answers to the following research questions:

1. Does breast cancer respond to Ispinesib?
2. What are the side effects of Ispinesib?
3. How much Ispinesib is in the blood at specific times after it is taken?

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB or Stage IV breast cancer
* Previously received anthracycline and taxane therapy

Exclusion criteria:

* Actively receiving anti-cancer therapy agent(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-06-30 (Actual); Primary Completion 2006-08-25 (Actual); Study Completion 2006-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (4):
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Pittsburgh, Pennsylvania
- GSK Investigational Site, Brussels, Belgium
- GSK Investigational Site, Bandar Tun Razak, Cheras, Malaysia
- GSK Investigational Site, Singapore, Singapore
- United Kingdom (4):
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Newcastle upon Tyne, Northumberland
  - GSK Investigational Site, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in females with advanced or metastatic breast cancer. The study was conducted from 30 January 2004 to 25 August 2006, with a total of 50 female participants enrolled in the study.
Groups:
- SB-715992: The eligible participants were administered Ispinesib, intravenously as a one-hour infusion on Day 1 of every 21-day treatment cycle, at a dose of 18 milligram (mg)/ meter square (m^2). The dosing was repeated for up to multiple cycles, until disease progression or removal from treatment due to an unacceptable toxicity or withdrawal of consent.
Period: Overall Study
Arm/Group | SB-715992
Started | 50
Completed | 0
Not Completed | 50
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Disease progression | 45
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- SB-715992: The eligible participants were administered Ispinesib, intravenously as a one-hour infusion on Day 1 of every 21-day treatment cycle, at a dose of 18 mg/m^2. The dosing was repeated for up to multiple cycles, until disease progression or removal from treatment due to an unacceptable toxicity or withdrawal of consent.
Arm/Group | SB-715992
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.7 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African heritage | 1
  Asian - Central/South Asian heritage | 2
  Asian - East Asian heritage | 6
  Asian - South East Asian heritage | 10
  White - Arabic/North African heritage | 1
  White - White/Caucasian/European heritage | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response Rate (ORR) Following Administration of Ispinesib
Description: Overall tumor response rate, was defined as the percentage of participants achieving either a complete response (CR) or partial response (PR), stable disease (SD), or progressive disease (PD). It was assessed by Computer tomography (CT) or Magnetic Resonance Imaging (MRI) scan. Response and progression was evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.0. The target lesions (TLs): CR, Disappearance of all TLs; PR where at least a 30% decrease in the sum of the longest diameter (LD) of TLs, taking as reference the baseline sum LD; PD : At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: After cycle 2 and repeated every 2 cycles up to Cycle 10, up to 26 months
Population: Intent to treat population consisted of all participants (n=50) who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SB-715992
Number analyzed (Participants) | 50
percentage of participants | 8

2. Secondary Outcome: Median Time to Response
Description: Time to response was defined as the time between the start of first dose of the study drug until the first documented evidence of partial or complete tumor response (whichever status was recorded first). When tumor response was confirmed at a repeat assessment, the time to response was taken as the first time the response was observed. For participants who did not show a tumor response, the time was censored at the time of withdrawal from the study for any reason. It was evaluated using RECIST criteria 1.0. CR for TLs was defined as Disappearance of all TLs and PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of TLs, taking as reference the baseline sum LD.
Time Frame: After cycle 2 and repeated every 2 cycles up to Cycle 10, up to 26 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | SB-715992
Number analyzed (Participants) | 50
weeks | 8.07 [5.4 to 10.7]

3. Secondary Outcome: Duration of Response
Description: For the participants who had a CR or PR, duration of response was defined as the time a CR or PR was first documented, until the first documented sign of disease progression or death. CR for TLs was defined as disappearance of all TLs and PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of TLs, taking as reference the baseline sum LD. The PD defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. For participants who did not progress or die, duration of response would be censored at the time of initiation of alternative anti-cancer therapy or time of last contact, if sooner. Due to small number of participants with a response, data was not summarized; however, individual participants data is reported week wise.
Time Frame: After cycle 2 and repeated every 2 cycles up to Cycle 10, up to 26 months
Population: ITT population. Only those participants available at that particular timepoints were analyzed
Measure: Number; unit: Weeks
Arm/Group | SB-715992
Number analyzed (Participants) | 4
Weeks
  Participant 1 | 6.9
  Participant 2 | 9
  Participant 3 | 11.7
  Participant 4 | 19.1

4. Secondary Outcome: Median Time-to-progression After Administration of Inspinesib
Description: Time-to-progression was defined as the time from the start of treatment until the first documented sign of disease progression or death due to any cause, if sooner. The PD as per RECIST criteria 1.0 was defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. For participants who did not progress or die, time-to-progression was censored at the time of initiation of alternative anti-cancer therapy or time of last contact, if sooner.
Time Frame: After cycle 2 and repeated every 2 cycles up to Cycle 10, up to 26 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: week
Arm/Group | SB-715992
Number analyzed (Participants) | 50
week | 5.86 [5.57 to 6.14]

5. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant.
Time Frame: From first dose of study drug (Day 1) to 30 days after the last dose (up to 26 months)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | SB-715992
Number analyzed (Participants) | 50
Participants
  Any SAEs | 23
  Any AE | 49
  Any deaths | 11

6. Secondary Outcome: Number of Participants With Clinical Concern Values for Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), Temperature and Heart Rate
Description: The vital sign examination included temperature, heart rate, SBP and DBP. Participant data for clinical concern vital parameters; SBP (unit: millimeter of Mercury [mmHg]: low concern (LC) and high concern (HC) values as 90 and 180 mmHg; DBP: LC and HC values as 40 and 100 mmHg; heart rate (units: beats per minute [bpm]): LC and HC as 50 and 140 bpm; and temperature (units: degree celsius): LC and HC as 36 and 41 degree Celsius; outside the mentioned range were reported. The available data for the participants from Cycle 1 (C1) Day 1 (D1); C2D1, C3D1, C4D1, C5D1, post-treatment and any visit post-screening were reported.
Time Frame: After cycle 2 and repeated every 2 cycles up to Cycle 10, up to 26 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | SB-715992
Number analyzed (Participants) | 50
Participants
  SBP, C1D1, Pre-dose, <CCR | 1
  SBP, C1D1, post-infusion, missing | 2
  SBP, C2D1, Missing | 1
  SBP, C5D1, Missing | 1
  SBP, post-treatment, Missing | 5
  SBP, any visit post-screen<CCR | 1
  DBP, C1D1, pre-dose, >CCR | 2
  DBP, C1D1, post-infusion, missing | 2
  DBP, C2D1, missing | 1
  DBP, C5D1, missing | 1
  DBP, post-treatment, Missing | 5
  DBP, post-treatment, >CCR | 2
  DBP, any visit post-screen, >CCR | 3
  HR, C1D1, post-infusion, Missing | 2
  HR, C2D1, Missing | 2
  HR, post-treament, Missing | 6
  Temperature, C1D1, pre-dose, Missing | 3
  Temperature, C1D1, pre-dose, < CCR | 3
  Temperature, C1D1, post-infusion, Missing | 7
  Temperature, C1D1, post-infusion, < CCR | 2
  Temperature, C2D1, Missing | 5
  Temperature, C2D1, < CCR | 4
  Temperature, C3D1, Missing | 1
  Temperature, C3D1, < CCR | 4
  Temperature, C4D1, Missing | 1
  Temperature, C4D1, < CCR | 2
  Temperature, C5D1, Missing | 1
  Temperature, post-treatment, Missing | 5
  Temperature, post-treatment, <CCR | 3
  Temperature, any visit post-screen, Missing | 2

7. Secondary Outcome: Number of Participants With Toxicity Shift Grade From Baseline for Hematology Parameters
Description: Blood samples for the assessment of hematology parameters were taken at intervals throughout the study. A total of 45 to 46 milliliter (ml) of blood over a 21-day cycle of treatment was collected. For hematology, the parameters assessed were: Hemoglobin, hematocrit, platelet count, Red blood cell count, white blood cell count (WBC), lymphocytes, monocytes, granulocytes, neutrophils, ,eosinophils and basophils. The toxicities for the hematology parameters were graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 3.0. Grade (G) 0= None (normal limits); G1= Mild, G2=Moderate; G3=Severe; G4= Fatal. The toxicity shift grades for Hemoglobin, Lymphocytes, Neutrophils, platelet count and WBC, were reported.
Time Frame: After cycle 2 and repeated every 2 cycles up to Cycle 10, up to 26 months
Population: ITT population. Only those participants with data available at the specified time points were analyzed (represented by n=X) in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | SB-715992
Number analyzed (Participants) | 50
Participants
  Hemoglobin, G0 to G1 | 12
  Hemoglobin, G0 to G2 | 4
  Hemoglobin, G1 to G2 | 8
  Hemoglobin, G1 to G4 | 1
  Lymphocytes, G0 to G1: number analyzed (Participants) | 49
  Lymphocytes, G0 to G1 | 3
  Lymphocytes, G0 to G2: number analyzed (Participants) | 49
  Lymphocytes, G0 to G2 | 4
  Lymphocytes, G0 to G3: number analyzed (Participants) | 49
  Lymphocytes, G0 to G3 | 2
  Lymphocytes, G1 to G2: number analyzed (Participants) | 49
  Lymphocytes, G1 to G2 | 7
  Lymphocytes, G1 to G3: number analyzed (Participants) | 49
  Lymphocytes, G1 to G3 | 1
  Lymphocytes, G1 to G4: number analyzed (Participants) | 49
  Lymphocytes, G1 to G4 | 1
  Lymphocytes, G2 to G3: number analyzed (Participants) | 49
  Lymphocytes, G2 to G3 | 3
  Neutrophils, G0 to G1 | 3
  Neutrophils, G0 to G2 | 6
  Neutrophils, G0 to G3 | 3
  Neutrophils, G0 to G4 | 26
  Neutrophils, G1 to G2 | 1
  Neutrophils, G1 to G3 | 1
  Neutrophils, G1 to G4 | 4
  Platelet count, G0 to G1 | 7
  Platelet count, G0 to G2 | 1
  WBC, G0 to G1 | 7
  WBC, G0 to G2 | 15
  WBC, G0 to G3 | 22
  WBC, G0 to G4 | 3
  WBC, G1 to G3 | 1
  WBC, G2 to G3 | 1
  WBC, G2 to G4 | 1

8. Secondary Outcome: Number of Participants With Toxicity Shift Grade From Baseline for Clinical Chemistry Grade Shifts
Description: Blood samples for the assessment of hematology parameters were taken at intervals throughout the study. A total of 45 to 46 milliliter (ml) of blood over a 21-day cycle of treatment was collected. For clinical chemistry, the parameters assessed were Alanine transaminase (ALT), Aspartate transaminase (AST), Hemoglobin, lymphocytes, neutrophils, platelet count, white blood cell (WBC), albumin, alkaline phosphatase increased, total bilirubin, calcium, creatinine, glucose, potassium and sodium. The toxicities for the clinical chemistry parameters were graded according to the NCI-CTCAE, version 3.0. where; G 0= None (normal limits); G1= Mild, G2=Moderate; G3=Severe; G4= Fatal. The number of participants with toxicity shift grades for clinical chemistry were reported.
Time Frame: After cycle 2 and repeated every 2 cycles up to Cycle 10, up to 26 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | SB-715992
Number analyzed (Participants) | 50
Participants
  ALT, G0 to G1 | 9
  ALT, G0 to G2 | 1
  ALT, G1 to G0 | 1
  ALT, G1 to G2 | 1
  ALT, G1 to G3 | 1
  ALT, G2 to G0 | 1
  AST, G0 to G1 | 14
  AST, G0 to G2 | 1
  AST, G1 to G0 | 1
  AST, G1 to G2 | 2
  AST, G1 to G3 | 2
  AST, G2 to G3 | 1
  Albumin, G0 to G1 | 7
  Albumin, G0 to G2 | 2
  Albumin, G1 to G0 | 3
  Albumin, G1 to G2 | 3
  Alkaline phosphatase, G0 to G1: number analyzed (Participants) | 49
  Alkaline phosphatase, G0 to G1 | 6
  Alkaline phosphatase, G1 to G2: number analyzed (Participants) | 49
  Alkaline phosphatase, G1 to G2 | 2
  Alkaline phosphatase, G1 to G3: number analyzed (Participants) | 49
  Alkaline phosphatase, G1 to G3 | 1
  Alkaline phosphatase, G2 to G1: number analyzed (Participants) | 49
  Alkaline phosphatase, G2 to G1 | 1
  Alkaline phosphatase, G2 to G3: number analyzed (Participants) | 49
  Alkaline phosphatase, G2 to G3 | 1
  Total Bilirubin, G0 to G1: number analyzed (Participants) | 49
  Total Bilirubin, G0 to G1 | 1
  Total Bilirubin, G0 to G4: number analyzed (Participants) | 49
  Total Bilirubin, G0 to G4 | 1
  Total Bilirubin, G1 to G3: number analyzed (Participants) | 49
  Total Bilirubin, G1 to G3 | 1
  Calcium, G0 to G1 | 9
  Calcium, G0 to G2 | 1
  Calcium, G1 to G4 | 1
  Creatinine, G0 to G1 | 3
  Glucose, G0 to G1 | 10
  Glucose, G0 to G2 | 1
  Glucose, G0 to G3 | 1
  Glucose, G1 to G0 | 2
  Glucose, G1 to G2 | 1
  Glucose, G1 to G3 | 1
  Glucose, G2 to G1 | 1
  Glucose, G2 to G3 | 1
  Glucose, G3 to G2 | 2
  Potassium, G0 to G1 | 11
  Sodium, G0 to G1 | 6
  Sodium, G0 to G3 | 3
  Sodium, G1 to G0 | 2
  Sodium, G1 to G3 | 1

9. Secondary Outcome: Pharmacokinetic (PK) Parameter-Clearance
Description: The assessment of clearance for SB-715992 was planned to be collected on C1D1 at timepoints; pre-dose, and post-dose 30 minute to 1 hour, 1.5 to 2.5 hours, 4 to 6 hours and 20 to 24 hours. However, the data for analysis of PK parameter was not collected.
Time Frame: Pre-dose, and post-dose 30 minute to 1 hour, 1.5 to 2.5 hours, 4 to 6 hours and 20 to 24 hours up to Cycle 10, up to 26 months
Population: The data for the outcome 'PK parameter-clearance' was not collected
Arm/Group | SB-715992
Number analyzed (Participants) | 0

10. Secondary Outcome: PK Parameter-Volume of Distribution
Description: The assessment of volume of distribution for SB-715992 was planned to be collected on C1D1 at timepoints; pre-dose, and post-dose 30 minute to 1 hour, 1.5 to 2.5 hours, 4 to 6 hours and 20 to 24 hours. Additional samples were to be collected in subsequent cycles, only if dose of study drug was adjusted for any reason following Cycle 1. However, the data for analysis of PK parameter was not collected.
Time Frame: as for outcome 9
Population: Data for PK parameter 'Volume of distribution' was not collected.
Arm/Group | SB-715992
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of first dose of study drug (D1) to 30 days after the last dose (Up to 26 months)
Description: ITT population was used for analysis.
Arm/Group | SB-715992
All-Cause Mortality (participants affected / at risk) | 11/50
Serious Adverse Events (participants affected / at risk) | 23/50
Other Adverse Events (participants affected / at risk) | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SB-715992 (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Pyrexia (General disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Catheter related infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SB-715992 (N=50)
Neutropenia (Blood and lymphatic system disorders) | 20
Vomiting (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.